CLINICAL TRIAL: NCT07111793
Title: IBSoFACTo : Identification of Clinical, Genetic and Immunological Factors Involved in the Development of Severe Bacterial Infections in Pediatrics
Brief Title: Identification of Clinical, Genetic and Immunological Factors Involved in the Development of Severe Bacterial Infections in Pediatrics
Acronym: IBSoFACTo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC25_0061; 2025-A01367-42 (Other: ANSM - IDRCB)
Record Dates: First submitted 2025-07-17; First posted 2025-08-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Severe Bacterial Infections
Keywords: Severe bacterial infections; Whole-exome sequencing; Inborn errors of immunity; pediatrics
MeSH Terms: conditions — Bacterial Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with severe childhood bacterial infections (Other): Patient inclus dans l'étude DIABACT IV (NCT02167802) entre 2015 et 2018, dans les suites de son hospitalisation en réanimation pédiatrique en France pour une infection bactérienne sévère.
  Interventions: Other: Extended phenotyping; Other: Blood sample for WES; Other: Blood sample for PBMC freezing; Other: POPC score evaluation; Other: Questionnaire completion
- Patient's biological parents (Other)
  Interventions: Other: Blood sample for WES; Other: Questionnaire completion

INTERVENTIONS:
Other: Extended phenotyping — Extended phenotyping (analysis performed at Nantes University Hospital, MANDATORY DELIVERY WITHIN 24 HOURS) = 1 EDTA 3 mL tube for patients included in Nantes.
  Arms: Patients with severe childhood bacterial infections
Other: Blood sample for WES — Blood sample for WES : 1 x 3 mL EDTA tube (if not included in DIABACT IV biocollection)
Other: Blood sample for PBMC freezing — Blood sample for PBMC freezing integrated into the biocollection: 1 EDTA tube = 3 mL
  Arms: Patients with severe childhood bacterial infections
Other: POPC score evaluation — Assessment of POPC score (Pediatric Overall Performance Category)
  Arms: Patients with severe childhood bacterial infections
Other: Questionnaire completion — Questionnaires completed by parents or children:
  * SDQ
  * PedSQL4.0

SUMMARY:
Severe bacterial infections (SBI) are responsible for significant morbidity and mortality in the paediatric population. There is considerable individual variability in children's susceptibility to developing SBIs. This variability is multifactorial, and the mechanisms at work are not yet fully understood. The investigators of this study therefore propose to study a population of children who had particularly severe bacterial infections requiring hospitalization in a pediatric intensive care unit in France between 2015 and 2018. This study is part of a global approach to understanding the mechanisms favoring the occurrence of IBS in pediatrics.

The study will initially focus on analyzing the clinical phenotype of these children in terms of the type of infection presented, as well as immunologically with an immune workup of all these patients. The investigators also plan to contact each family individually to identify other episodes of personal or family IBS or other elements suggestive of immune deficiency (opportunistic infections, autoimmune manifestations, severe atopy). The investigators will also assess the persistent sequelae since their infectious episode, and their quality of life following this IBS.

In parallel, the genetic analysis of these patients and their parents will be carried out using whole-exome sequencing. The investigators will compare the results with those obtained in 2 IBS-free control populations (N=70 and N=116). The goal is to identify genetic variants that favor the occurrence of IBS in general, and some that are specific to certain bacteria or clinical presentations.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Patient included in the DIABACT IV study between 2015 and 2018, following hospitalization in a pediatric intensive care unit in France for a severe bacterial infection.
* Patient affiliated to a social security system
* Patient alive at the time of inclusion.
* Written consent from legal representatives for participation in research. If one of the legal representatives is unable to complete/sign the written consent, it will be sought orally by telephone and recorded in the patient's file. If the patient is over 18, written consent will be obtained. If the patient is a minor, consent will be sought with communication adapted to his/her level of understanding and age.

For parents:

* Patient's biological parents
* Written consent

Exclusion Criteria:

* Persons under court protection
* Refusal to participate in research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1401 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of innate errors of immunity involved in the development of IBS in pediatrics. | At the enrollment
  List of rare genetic variants significantly more frequently found in cases than in controls and/or absent in healthy parents.

SECONDARY OUTCOMES:
Identification of inborn errors of immunity involved in the development of IBS and their association with abnormalities of the immune balance, | At the enrollment
Identification of rare genetic variants favoring certain clinical types of infection, or certain biological and immunological abnormalities. | At the enrollment
Identification of immune deficiencies in patients who have developed a severe bacterial infection | At the enrollment
Assessment of sequelae with the POPC sequelae score (Pediatric Overall Performance Category) at a distance from the IBS episode. | At the enrollment
  The POPC sequelae score is a scale from 1 to 6, with 6 being the worst possible outcome.
Assessment of sequelae at a distance from the IBS episode with the Strengths and Weaknesses Questionnaire (SDQ-Fra). | At the enrollment
  The SDQ-Fra score is a scale from 0 to 2, with 2 being the worst possible outcome.
Assessment of quality of life at a distance from the IBS episode. | At the enrollment
  Quality of life will be assessed in this patient population using the Pediatric Quality of Life InventoryTM (scale from 0 to 4, with 4 corresponding to the worst outcome).

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Nantes University Hospital, Nantes, Loire Atlantique
  - CHU de Brest, Brest
  - Hospices Civils de Lyon, Lyon
  - Hôpital Armand Trousseau, Paris
  - Hôpital Necker enfants malades, Paris
  - CHU de Saint-Étienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided